CLINICAL TRIAL: NCT03319745
Title: A Window of Opportunity Phase II Study of Pembrolizumab in Patients With Bladder Cancer Undergoing Radical Cystectomy
Brief Title: Pembrolizumab in Treating Patients With Bladder Cancer Undergoing Radical Cystectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0057; NCI-2018-01032 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0057 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-10-20; First posted 2017-10-24 (Actual); Results first posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Stage I Bladder Cancer AJCC v8; Stage II Bladder Cancer AJCC v8; Stage III Bladder Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8; Stage IIIB Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 2 cycles in the absence of disease progression or unacceptable toxicity. About 4 weeks after treatment, patients then undergo radical cystectomy per standard of care.
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies the side effects of pembrolizumab and to see how well it works in treating patients with bladder cancer who are undergoing surgery to remove the bladder. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To characterize the safety profile of pembrolizumab in patients with urothelial carcinoma undergoing radical cystectomy.

SECONDARY OBJECTIVES:

I. To explore a signal of anti-cancer immunological activity by evaluating surgical specimens for evidence of post-treatment lymphocytic infiltration and residual tumor compared to pre-treatment biopsy samples.

II. To explore a signal of biomarker activity by evaluating surgical specimens and blood samples for established and not-so-established markers of response to pembrolizumab.

III. To report the tumor yield and sufficiency of tumor for immunological and biomarker activity.

IV. To examine the interaction of the human microbiome and pathologic response to pembrolizumab.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 2 cycles in the absence of disease progression or unacceptable toxicity. About 4 weeks after treatment, patients then undergo radical cystectomy per standard of care.

After completion of study treatment, patients are followed up to 30 and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent.
* Have absence of metastatic disease as determined by conventional imaging studies and be considered a good surgical candidate by the treating physician.
* Be willing to participate in the collection of blood and tissue for banking and future correlative studies.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale.
* Absolute neutrophil count (ANC) >= 1,500 /mcL.
* Platelets >= 100,000/mcL.
* Hemoglobin (Hgb) >= 9 g/dL or >= 5.6 mmol/L without (w/o) transfusion within 7 days of assessment.
* Creatinine OR calculated creatinine clearance =< 1.5 x upper limit of normal (ULN) OR >= 30 mL/min for subject with creatinine levels > 1.5 x institutional ULN. Creatinine clearance should be calculated per institutional standard.
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 x ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN OR =< 5 x ULN for subjects with liver metastases.
* Albumin > 2.5 mg/dL.
* Coagulation international normalized ratio (INR) or prothrombin time (PT) activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Male subjects of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Is currently participating and receiving pembrolizumab or has participated in a study of an investigational agent and received pembrolizumab or used an investigational device within 4 weeks of the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Has a known history of active TB (Bacillus tuberculosis).
* Has a known history of hypersensitivity to pembrolizumab or any of its excipients.
* Has had prior systemic anti-cancer therapy for the treatment of bladder cancer. Prior intravesical therapies, whether Bacillus Calmette-Guerin (BCG) (including but not limited to: persistent high-grade disease or recurrence within 6 months of receiving at least two courses of intravesical BCG [at least five of six induction doses and at least two of three maintenance doses]; or T1 high-grade disease at the first evaluation following induction BCG alone [at least five of six induction doses]), chemotherapy or otherwise, will remain eligible.
* Has any other malignancy diagnosed within 2 years of screening with the exception of basal or squamous cell skin cancer, or non-invasive cancer of the cervix, or any other cancer deemed by the treating physician to be of low-risk for progression or patient morbidity during the study period.
* Has known metastatic disease as determined by conventional staging studies.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has a clinically significant active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating physician.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected).
* Has received a live vaccine within 30 days of initiation of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neema Navai, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 participants consented, 6 screen failed. 18 participants were found eligible to receive study treatment. 16 out of the 18 were able to undergo surgery.
Groups:
- Pembrolizumab: Participants receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 2 cycles in the absence of disease progression or unacceptable toxicity. About 4 weeks after treatment, participants then undergo radical cystectomy per standard of care.
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 18
Completed | 16
Not Completed | 2
Not completed — Death | 1
Not completed — Toxicity Precluding Surgery | 1

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 2 cycles in the absence of disease progression or unacceptable toxicity. About 4 weeks after treatment, patients then undergo radical cystectomy per standard of care.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Toxicity for Safety Monitoring (TOX)
Description: The primary endpoint is a joint endpoint classifying patients as having a toxicity of concern (TOX), defined as the presence of any of these: 1) any 30-day grade 3 or higher surgical complication at least possibly related to the treatment, 2) any toxicity at least possibly related to the treatment that prevents surgery, or 3) death between the start of the study and the 30-day post-surgical assessment as long as it is at least possibly related to pembrolizumab or surgery.
Time Frame: From initiation of pembrolizumab, until 90 days post-surgery, up to a maximum of 5.5 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 18
percentage of participants | 15 [3 to 33]

2. Secondary Outcome: Efficacy Endpoint
Description: To explore anti-cancer immunological activity by evaluating surgical specimens for evidence of post-treatment and residual tumor compared to pre-treatment biopsy samples. The main mechanism for doing so will be via histopathologic review of the radical cystectomy specimen. MIBC participants are defined as responders if they achieve a pT1 stage or less. In the case of NMIBC a pT0 status will be used to identify complete response.
Time Frame: Efficacy endpoint will be measured at time of surgery
Population: Only 16 participants were included in the analysis of this outcome as 2 of the 18 participants were unable to undergo surgery; therefore, we did not have their surgical specimens.
Measure: Number; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 16
Participants | 5

ADVERSE EVENTS:
Time Frame: From initiation of pembrolizumab, until 90 days post-surgery, up to a maximum of 5.5 months
Description: From the time of initiation of pembrolizumab through 30 days after surgery, all adverse events must be reported by the investigator. Additionally, all adverse events meeting serious criteria, from time of treatment initiation through 90 days following cessation of study treatment, or 30 days following cessation of study treatment if the participant initiates new anti cancer therapy should be reported by the investigator.
Arm/Group | Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 9/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=18)
Sepsis (Infections and infestations) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Thromboemolic Event (Vascular disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Small Intestinal Leak (Gastrointestinal disorders) | 1 (1)
Acute Pyelonephritis (Renal and urinary disorders) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Enterocolitis Infectious (Infections and infestations) | 1 (1)
Pelvic Infection (Infections and infestations) | 2 (2)
UTI (Renal and urinary disorders) | 2 (2)
Ureteric Anastomotic Leak (Renal and urinary disorders) | 1 (1)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=18)
Anemia (Blood and lymphatic system disorders) | 14 (14)
Fatigue (General disorders) | 9 (9)
Hyponatremia (Investigations) | 7 (7)
Creatinine Increased (Renal and urinary disorders) | 4 (4)
Hypokalemia (Investigations) | 3 (3)
ALT Increased (Investigations) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Nausea/Vomiting (Gastrointestinal disorders) | 3 (3)
UTI (Renal and urinary disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
ALK Increased (Investigations) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 2 (2)
Lipase Increased (Investigations) | 2 (2)
Tachicardia (Cardiac disorders) | 2 (2)
Platelet Count Decreased (Blood and lymphatic system disorders) | 2 (2)
AST Increased (Investigations) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Dematitis (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
WBC Decreased (Blood and lymphatic system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Anxiety (Nervous system disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Weakness (Nervous system disorders) | 1 (1)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperuricemia (Investigations) | 1 (1)
Hypermagnesemia (Investigations) | 1 (1)
Hyperkalemia (Investigations) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Hot Flashes (General disorders) | 1 (1)
Stoma Infection (Infections and infestations) | 1 (1)
Edema Limbs (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT03319745/Prot_SAP_000.pdf